CLINICAL TRIAL: NCT03086044
Title: Transplanting Organs From Hepatitis C Positive Donors to Hepatitis C Uninfected Recipients
Brief Title: Transplanting Hepatitis C Positive Organs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lindsey R. Baden, MD, Associate Professor at Harvard Medical School, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-P001170
Record Dates: First submitted 2016-09-12; First posted 2017-03-22 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Hepatitis C; Awaiting Organ Transplant
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; Sofosbuvir; velpatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCV NAT Positive Donor (Experimental): Intervention: 2 week treatment course with a direct acting antiviral, sofosbuvir 400mg / velpatasvir 100mg daily
  Participants who receive allografts from a donor who is HCV NAT positive will receive treatment with a direct acting antiviral, sofosbuvir 400mg / velpatasvir 100mg daily, beginning on the day of transplant.
  Interventions: Drug: Sofosbuvir/velpatasvir
- HCV NAT Negative, HCV Ab Positive Donor (Experimental): Intervention: HCV viral load monitoring
  Participants who receive allografts from a donor who is HCV Ab positive and NAT negative will have close serial HCV viral load monitoring and will be treated with a direct acting antiviral, 400mg / velpatasvir 100mg daily, for 6 weeks if HCV viremia develops.
  Interventions: Drug: Sofosbuvir/velpatasvir; Other: Monitoring

INTERVENTIONS:
Drug: Sofosbuvir/velpatasvir — 2 weeks of treatment beginning on the day of transplant
  Other Names: Epclusa
Other: Monitoring — Close HCV viral load monitoring Will receive direct acting antiviral treatment with 6 weeks of sofosbuvir/velpatasvir if the recipient develops HCV viremia during the post-transplant HCV viral load testing
  Other Names: Sofosbuvir/velpatasvir (Epclusa)
  Arms: HCV NAT Negative, HCV Ab Positive Donor

SUMMARY:
This is an open-label, pilot safety and efficacy trial for adults who are active on the heart, lung, or kidney transplantation lists and are eligible to receive an organ from an increased risk donor who has evidence of active or prior hepatitis C infection (HCV).

DETAILED DESCRIPTION:
This is an open label pilot study transplanting organs from Hepatitis C positive donors into HCV uninfected recipients at Brigham and Women's Hospital. Heart, lung and kidney transplant participants will be stratified into two different study arms depending on whether the donor of the organ was HCV nucleic acid amplifications technology (NAT) positive or negative. In the NAT positive arm, the recipients will receive a course of direct acting antivirals (DAA) to begin on the day of transplant. If the donor was HCV antibody (Ab) positive and NAT negative, the recipients will receive close monitoring with serial HCV viral loads (VL) and will only begin treatment with DAA if they develop HCV viremia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are age ≥ 18 years
* Active on either the cardiac, lung, or kidney transplant waiting list
* Willing and able to provide written informed consent to receive organs from an increased risk donor with a known transmissible infection

Exclusion Criteria:

* Hepatitis B NAT or viral load positive
* Evidence of cirrhosis or clinically significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Graft survival | 6 months post-transplant
  Functioning allograft not requiring mechanical support
HCV status of the transplant recipient | 6 months post-transplant
  Sustained virologic response (SVR) 12 weeks after HCV treatment completion in Arm A or at 6 months in Arm B (SVR defined as HCV RNA < lower limit of quantification)

SECONDARY OUTCOMES:
Treatment related adverse events | 6 months post-transplant
  Number of treatment related adverse events per patient using direct-acting antiviral HCV regimens in post transplant recipients

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woolley AE, Singh SK, Goldberg HJ, Mallidi HR, Givertz MM, Mehra MR, Coppolino A, Kusztos AE, Johnson ME, Chen K, Haddad EA, Fanikos J, Harrington DP, Camp PC, Baden LR; DONATE HCV Trial Team. Heart and Lung Transplants from HCV-Infected Donors to Uninfected Recipients. N Engl J Med. 2019 Apr 25;380(17):1606-1617. doi: 10.1056/NEJMoa1812406. Epub 2019 Apr 3. PMID 30946553